CLINICAL TRIAL: NCT02090998
Title: A Comparison of the Efficacy of 5% Lidocaine Anesthetic to Provide SPGB Vs. Elavil for the Treatment of Transformed Migraine
Brief Title: Sphenopalatine Ganglion Nerve Block vs. Elavil for Treatment of Transformed Migraines
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: no patients during covid pandemic
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, William Grubb, M.D., Associate Prof., Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2012002610
Record Dates: First submitted 2014-03-17; First posted 2014-03-19 (Estimated); Results first posted 2021-12-29 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2023-05

CONDITIONS: Transformed Migraine; Chronic Daily Headache
Keywords: Migraine Headache; Menstrual Migraine; Vascular Headache; Temporal Lobe Seizure
MeSH Terms: conditions — Headache Disorders; Migraine Disorders; Vascular Headaches; Epilepsy, Temporal Lobe | interventions — Amitriptyline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SPG Nerve Block with Lidocaine 5% gel (Active Comparator): Sphenopalatine Ganglion Nerve Block (SPG Nerve Block) will be administed weekly for 4 weeks using 5% Lidocaine gel This intervention (a nerve block) will treat the headache for the time period investigated
  Interventions: Procedure: SPG Block with 5% Lidocaine gel; Drug: Amitriptyline
- Amitriptyline / Elavil (Active Comparator): Amitriptyline / Elavil 10 mg once a day for one week then Amitriotyline 20 mg once a day for three weeks This intervention will treat the headache for the time period investigated
  Interventions: Procedure: SPG Block with 5% Lidocaine gel; Drug: Amitriptyline

INTERVENTIONS:
Procedure: SPG Block with 5% Lidocaine gel — cotten tipped applicators are with 5% lidocaine gel and placed in the nares to lye in the skin over the sphenopalitine ganglion. The applcator is use to saturate the spenopalitine ganglion with 5ml of 1% lidocaine local anesthesia
Drug: Amitriptyline — The intervention will be Amitriptyline daily (starting with 10 mg) PO for 30 Days
  Other Names: Elavil

SUMMARY:
This study will compare a local anesthetic technique that has been used to treat subjects suffering from transformed migraines (chronic migraines) versus medical management with traditional antidepressant Amitriptyline / Elavil.

Subjects will be randomized into one of two treatment groups to compare the safety and efficacy of the therapies. Subjects will recieve either sphenopalatine ganglion nerve block with 5% lidocaine gel into the nasopharynx or medical management with traditional antidepressants, Elavil, to produce a reduction in the frequency and severity of the headache.

We propose that there will be a difference in the outcomes when comparing the two methods of treating transformed migraines and that one research arm will result in more patient satisfaction and greater efficacy in the treatment of subjects

DETAILED DESCRIPTION:
Arm one will receive Sphenopalatine Ganglion Nerve Block weekly for 4 weeks

Arm two will receive Amitriptyline / Elavil daily for 30 Days

ELIGIBILITY:
Inclusion Criteria:

1. Male and female age 18-90
2. Subject have formal medical diagnosis of migraine headache
3. Subjects currently require treatment for headache
4. Subjects who have received optimal medical management from migraines including triptans (Imitrex, Amerge and Relpax)
5. Subjects who have recieved optimal medical management for migraines including anticonvulsants (Depakote, Lamictal, klonopin

Exclusion Criteria:

1. Less than 18 years of age
2. Subjects will be excluded if they are already being treated with lidocaine (patch or other vehicle) for chronic pain
3. Untreated Heart Failure
4. Pregnancy
5. Individuals unwilling to comply with study procedures and follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-05; Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rutgers, Robert Wood Johnson Medical School , Pain Center of NJ, New Brunswick, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Amitriptyline / Elavil | SPG Nerve Block With Lidocaine 5% Gel
Started | 2 | 8
Completed | 2 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amitriptyline / Elavil | SPG Nerve Block With Lidocaine 5% Gel | Total
Number analyzed (Participants) | 2 | 8 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 8 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 46 [45 to 48] | 59 [39 to 84] | 56 [39 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 0 | 3 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 8 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 8 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 8 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Daily Headaches
Description: The number of times per day that symptoms occur
Time Frame: Study Day 1 through Study Day 30
Population: participants from 18-82 who had failed conventional headache therapies
Measure: Mean (Standard Deviation); unit: Number of Daily Headaches
Groups:
- Amitriptyline / Elavil: Amitriptyline / Elavil 10 mg once a day for one week then Amitriotyline 20 mg once a day for three weeks This intervention will treat the headache for the time period investigated SPG Block with 5% Lidocaine gel: cotten tipped applicators are with 5% lidocaine gel and placed in the nares to lye in the skin over the sphenopalitine ganglion. The applcator is use to saturate the spenopalitine ganglion with 5ml of 1% lidocaine local anesthesia
  Amitriptyline: The intervention will be Amitriptyline daily (starting with 10 mg) PO for 30 Days
Arm/Group | Amitriptyline / Elavil | SPG Nerve Block With Lidocaine 5% Gel
Number analyzed (Participants) | 2 | 8
Number of Daily Headaches | 20.5 (0.5) | 13.4 (10.4)

2. Other Pre Specified Outcome: Duration of Inactivity Associated With Headaches
Description: The time after events that effects patient activity level
Time Frame: Study Day 1 thorugh Study Day 30
Reporting Status: Not Posted

3. Post Hoc Outcome: Length of Duration of Headache
Description: Length of Duration of Headache
Time Frame: Greater than 20 minutes
Reporting Status: Not Posted, anticipated posting 2024-12

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Amitriptyline / Elavil | SPG Nerve Block With Lidocaine 5% Gel
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/8
Other Adverse Events (participants affected / at risk) | 0/2 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/98/NCT02090998/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/98/NCT02090998/ICF_001.pdf